CLINICAL TRIAL: NCT02568176
Title: An Open-Label Study to Evaluate the Pharmacokinetics of Intranasal Esketamine and Its Effects on the Pharmacokinetics of Orally-Administered Midazolam and Bupropion in Healthy Subjects
Brief Title: Pharmacokinetic Study of Intranasal Esketamine and Its Effects on the Pharmacokinetics of Orally-Administered Midazolam and Bupropion in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108043; ESKETINTRD1010 (Other: Janssen Research & Development, LLC); 2015-002654-13 (EudraCT Number)
Record Dates: First submitted 2015-10-02; First posted 2015-10-05 (Estimated); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Healthy
Keywords: Healthy; Pharmacokinetics; Esketamine; JNJ-54135419; Midazolam; Bupropion
MeSH Terms: interventions — Midazolam; Esketamine; Bupropion

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cohort 1 (Experimental): Participants will receive single oral dose of midazolam 6 milligram (mg) on Day 1 and 17. Participants will self-administer esketamine intranasally thrice per day on morning of Day 2, 5, 9, 12 and 16 (84 mg).
  Interventions: Drug: Midazolam; Drug: Esketamine
- Cohort 2 (Experimental): Participants will receive single oral dose of bupropion 150 mg on Day 1 and 19. Participants will self-administer esketamine intranasally thrice per day on morning of Day 4, 7, 11, 14 and 18 (84 mg).
  Interventions: Drug: Esketamine; Drug: Bupropion

INTERVENTIONS:
Drug: Midazolam — Single oral dose of midazolam 6 mg Day 1 and Day 17.
  Arms: Cohort 1
Drug: Esketamine — Intranasal esketamine will be self-administered 5 times during 15 days.
  Other Names: JNJ-54135419
Drug: Bupropion — Single oral dose of bupropion 150 mg on Day 1 and 19.
  Arms: Cohort 2

SUMMARY:
The primary purpose of this study is to evaluate the induction potential of repeated administration of intranasal esketamine on cytochrome P450 (CYP) 3A4 and CYP2B6 activity in healthy participants using orally administered midazolam and bupropion as probes, respectively and to evaluate the pharmacokinetics of esketamine after a single dose and repeated administration.

DETAILED DESCRIPTION:
This is a parallel group, single-center, repeat-dose, fixed-sequence, open-label (all people know the identity of the intervention), study. The effects of repeated administration of intranasal esketamine on the pharmacokinetics of midazolam and bupropion will be evaluated in Cohort 1 and Cohort 2, respectively. Participants in Cohort 1 will receive a single oral dose of midazolam in the morning of Day 1 and Day 17. Participants in Cohort 2 will receive a single oral dose of bupropion in the morning of Day 1 and Day 19. In Cohort 1 and 2 participants will self-administer 5 doses of intranasal esketamine over a 15-day period. The duration of study, from the Screening Phase through Follow-up, is up to 51 days and 54 days for Cohort 1 and Cohort 2, respectively. Blood samples for participants in Cohort 1 will be collected for up to 24 hours after dosing on Days 1 and 17 (midazolam) and for up to 24 hours on Days 2 and 16 (esketamine); For participants in Cohort 2, blood and urine samples for assessment of bupropion pharmacokinetics will be collected for up to 72 hours after dosing on Day 1 and Day 19. Participants' safety will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Be a man or woman of non-Asian origin 18 to 55 years of age, inclusive
* Signed an informed consent document indicating they understand the purpose of and procedures required for the study and are willing to participate in the study
* A woman of child-bearing potential, must have a negative serum β-human chorionic gonadotropin (hCG) pregnancy test at Screening and a negative urine pregnancy test on Day -1 of the treatment period. Women using contraceptives must agree to use an additional birth control method during the study and for 1 month after receiving the last dose of study drug
* A man who is sexually active with a woman of childbearing potential and has not had a vasectomy, must agree to use an adequate contraception method as deemed appropriate by the investigator (eg, vasectomy, double-barrier, partner using effective contraception) and to not donate sperm during the study and for 3 months after receiving the last dose of study drug
* Comfortable with self-administration of intranasal medication and able to follow instructions provided

Exclusion Criteria:

* Clinically significant abnormal values for hematology, clinical chemistry (particularly potassium or magnesium levels below the normal laboratory range), or urinalysis at Screening or at admission to the study center (Day -1) as deemed appropriate by the investigator
* Clinically significant abnormal physical examination, vital signs, or 12 lead electrocardiogram (ECG) at Screening or at admission to the study center (Day -1) as deemed appropriate by the investigator
* Use of any prescription or non-prescription medication (including vitamins and herbal supplements), except for paracetamol, contraceptives, and hormonal replacement therapy, within 14 days before the first dose of the study drug is scheduled until completion of the study
* Has used nasal tobacco powder ("snuff") regularly within the past year.
* Has a nasal piercing

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 71 (Actual)
Dates: Start 2015-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Maximum Plasma Concentration (Cmax) | up to Day 17 for Cohort 1; up to Day 19 for Cohort 2
  The Cmax is the maximum plasma concentration.
Time to reach maximum concentration (tmax) | up to Day 17 for Cohort 1; up to Day 19 for Cohort 2
  Time to reach the maximum observed plasma concentration.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-infinity]) | up to Day 17 for Cohort 1; up to Day 19 for Cohort 2
  The AUC (0-infinity) is the area under the plasma concentration-time curve from time zero to infinite time, calculated as the sum of AUC(last) and C(last)/lambda(z), wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time; and C(last) is the last observed quantifiable concentration; and lambda(z) is elimination rate constant.
Area Under the Plasma Concentration-Time Curve From Time Zero to Infinite Time (AUC [0-last]) | up to Day 17 for Cohort 1; up to Day 19 for Cohort 2
  The AUC (0-last) is the area under the plasma concentration-time curve from time zero to last quantifiable time, calculated as the sum of AUC(last) and C(last)/lambda(z), wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time; and C(last) is the last observed quantifiable concentration; and lambda(z) is elimination rate constant.
Terminal Half-Life(t[1/2]) | up to Day 17 for Cohort 1; up to Day 19 for Cohort 2
  Terminal half-life (t[(1/2]) is defined as 0.693/Lambda(z).
Area Under the Plasma Concentration-Time Curve From Time Zero to 12 hours (AUC [0-12]) | up to Day 17 for Cohort 1; up to Day 19 for Cohort 2
  The AUC (0-12) is the area under the plasma concentration-time curve from time zero to 12 hours, calculated as the sum of AUC(last) and C(last)/lambda(z), wherein AUC(last) is area under the plasma concentration-time curve from time zero to last quantifiable time; and C(last) is the last observed quantifiable concentration; and lambda(z) is elimination rate constant.
Cmax metabolite to parent ratio (MPR Cmax) | up to Day 17 for Cohort 1; up to Day 19 for Cohort 2
  Cmax metabolite to parent ratio, and corrected for molecular weight if necessary.
AUC(last) metabolite to parent ratio (MPR AUC[last]) | up to Day 17 for Cohort 1; up to Day 19 for Cohort 2
  AUC(last) metabolite to parent ratio, and corrected for molecular weight if necessary.
AUC (infinity) metabolite to parent ratio (MPR AUC [infinity]) | up to Day 17 for Cohort 1; up to Day 19 for Cohort 2
  AUC (infinity) metabolite to parent ratio, and corrected for molecular weight if necessary.
Amount of Drug excreted in Urine (Ae) | up to Day 17 for Cohort 1; up to Day 19 for Cohort 2
  Total amount excreted into the urine, calculated as the sum of all Ae(t1-t2) intervals.
Percentage of Drug dose excreted into urine | up to Day 19 for Cohort 2
  Total amount excreted into the urine, expressed as a percentage of the administered dose, calculated as (Ae/dose)*100, and corrected for molecular weight if necessary.
Renal clearance | up to Day 19 for Cohort 2
  Renal clearance calculated as Ae/AUC (infinity).
Formation Clearance | up to Day 19 for Cohort 2
  Formation clearance of drug, calculated as Ae of hydroxybupropion/AUC(infinity) of bupropion, and corrected for molecular weight if necessary.
Ae metabolite to parent ratio (MPR Ae) | up to Day 19 for Cohort 2
  Ae metabolite to parent ratio, and corrected for molecular weight if necessary.

SECONDARY OUTCOMES:
Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs) | Baseline up to Day 51 for Cohort 1; Baseline up to Day 54 Cohort 2
  An AE was any untoward medical event that occurs in a participant administered an investigational product, and it does not necessarily indicate only events with clear causal relationship with the relevant investigational product. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged in-patient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Merksem, Belgium

REFERENCES:
- [Derived] Perez-Ruixo C, Rossenu S, Zannikos P, Nandy P, Singh J, Drevets WC, Perez-Ruixo JJ. Population Pharmacokinetics of Esketamine Nasal Spray and its Metabolite Noresketamine in Healthy Subjects and Patients with Treatment-Resistant Depression. Clin Pharmacokinet. 2021 Apr;60(4):501-516. doi: 10.1007/s40262-020-00953-4. Epub 2020 Oct 31. PMID 33128208